CLINICAL TRIAL: NCT05101850
Title: Measurement of the Metabolic Cost of Inspiratory Muscle Training and Physical Rehabilitation in Mechanically Ventilated Patients; a Feasibility Study
Brief Title: Metabolic Cost of IMT
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Other Study IDs: 298839
Record Dates: First submitted 2021-09-30; First posted 2021-11-01 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mechanical ventilation is a life-saving intervention used worldwide. Despite this, critically ill patients who undergo mechanical ventilation commonly develop muscle weakness; this includes limb muscle weakness and diaphragmatic weakness.

Physiotherapy interventions on critically ill patients include; mobilisation to improve limb muscle strength and function, and inspiratory muscle training which aims to target the diaphragm and accessory inspiratory muscles with the goal of improving endurance and strength. Whilst these interventions are standard practice in intensive care, little is known about the physiological load imposed on patients.

The purpose of this study is to assess the feasibility of using indirect calorimetry (measured using the Beacon Caresystem) to measure the metabolic cost (oxygen consumption [VO2] and carbon dioxide production [VCO2]) of inspiratory muscle training and physical rehabilitation in mechanically ventilated intensive care patients.

DETAILED DESCRIPTION:
This is an initial cross-sectional study using a non-randomised convenience sample. Patients will be studied during either rehabilitation or Inspiratory Muscle Training.

All participants will have Maximal Inspiratory Pressure (PImax) measured every 5 days. Baseline measurements of VO2 and VCO2 at rest on their baseline ventilation will be measured using the Beacon Caresystem for 1 hour before Inspiratory Muscle Training or physical rehabilitation is initiated.

Inspiratory muscle training will will performed using a resistive device (Philips Respironics ® Threshold PEP device) which is inserted into the participants ventilator tubing 30 minutes before starting inspiratory muscle training. At this point, the device will be set to its lowest setting; the resistance will be overcome by support delivered through the ventilator meaning no additional effort for the participant.

The patient will then perform 12 breaths of inspiratory muscle training at 4cmH20, and at 30%, 50% and 80% PImax with a 30 second rest every 6 breaths and a 10-20 minute rest every 12 breaths

Inspiratory muscle training will normally occur five days per a week. The Beacon Caresystem will be connected for analysis up to 2 days per week.

Participants will receive usual physiotherapy exercise. These will be prescribed by the patient's physiotherapist and may include assisted mobilisation and / or upper and lower limb exercises to help strengthen muscles. Exercises performed will be categorised for analysis in the study according to a scale called the intensive care mobility scale.

When physical rehabilitation begins (i.e when the patient starts to move with the physiotherapist); a time stamp will be activated on the Beacon Caresystem. When physical rehabilitation has ended the time stamp will be deactivated.

Immediately after exercise the patient will be asked to rate their exertion using a simple scale designed to measure physical effort, called the BORG rating scale of perceived exertion.

Physical rehabilitation will normally occur six days per a week. The Beacon Caresystem will be connected for analysis up to 4 days per week.

ELIGIBILITY:
Inclusion Criteria:

* Patient invasively ventilated for ≥ 72 hours
* Have an endotracheal tube or tracheostomy in situ
* Respiratory rate of ≤ 35 breaths/min
* Fraction Inspired Oxygen (Fi02) ≤ 0.50
* Co-operative and able to participate in physical rehabilitation and inspiratory muscle training
* Age ≥ 18 years
* Patient consent or, in the case that the patient is unable, advice from the next of kin and acceptance of oral and written information describing the study.

Exclusion Criteria:

* Undrained pneumothorax/pneumomediastinum
* The absence of an arterial catheter for blood sampling at study start
* Unlikely to survive
* Pregnancy
* Consultant discretion that patient is not appropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Recruitment | Through study completion, 9 months
  The number of patients recruited to the trial compared to the number of eligible patients within the recruitment window
Adherence to IMT | Throughout the trial period of each participant whilst enrolled i study
  The adherence to the prescribed IMT protocol, including reasons for non-adherence
Prevalence of technical issues with relation to the Beacon Caresystem | Through study completion, 9 months
  Defined as inability to calibrate before intervention, missing data during interventions, inability to analyse data from interventions.

SECONDARY OUTCOMES:
Assessment of VO2 and VCO2 in ICU patients at rest | 60 minutes before physical rehabilitation or inspiratory muscle training
  Measured in ml/kg/min calculated as the mean VO2 and VCO2 during 60 consecutive minutes where there was a <10% variation in VO2 and VCO2 at rest
Comparison of VO2 and VCO2 during IMT at different percentages of PImax within and between patients | During inspiratory muscle training and for 30 minutes after inspiratory muscle training has ceased
  Measured in ml/kg/min for the total IMT session (2 sets of 6 breaths) and 30 minutes after the intervention (analysis of recovery time to baseline)
Prevalence of low PImax in patients receiving mechanical ventilation and PImax change during course of their admission | Day 0 (baseline) and every 5 days whilst the participant is enrolled in the study
  Measured in cmH20 at baseline and every five days
Comparison of VO2 and VCO2 during physical rehabilitation in patients receiving mechanical ventilation | During physical rehabilitation and for 30 minutes after physical rehabilitation has ceased
  Measured in ml/kg/min 30 minutes before the intervention, total VO2 and VCO2 during the intervention and 30 minutes after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Micheal Polkey, PhD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- The Royal Brompton and Harefield Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jenkins TO, Karbing DS, Rees SE, Poulsen MK, Patel BV, Polkey MI, MacBean V. Metabolic cost of physical rehabilitation in mechanically ventilated patients in critical care: an observational study. BMJ Open Respir Res. 2025 Apr 5;12(1):e002878. doi: 10.1136/bmjresp-2024-002878. PMID 40187744
- [Derived] Jenkins TO, MacBean V, Poulsen MK, Karbing DS, Rees SE, Patel BV, Polkey MI. The metabolic cost of inspiratory muscle training in mechanically ventilated patients in critical care. Intensive Care Med Exp. 2023 Jul 7;11(1):41. doi: 10.1186/s40635-023-00522-6. PMID 37415048